CLINICAL TRIAL: NCT04902898
Title: Evaluation of the Safety and Efficacy of the Sterile Single-use Circular Stapling Device CIRCCURER II (Jiangxi Langhe Medical Instrument Co., Ltd., Guangzhou, China) in Adult Patients Suffering From Pathologic Foreskin (Phimosis, Stenosis, Redundant Prepuce): A Prospective Randomised Comparative Clinical Trial
Brief Title: Safety and Efficacy of the Sterile Single-use Circular Stapling Device CIRCCURER II (Jiangxi Langhe Medical Instrument Co., Ltd., Guangzhou, China)
Acronym: CiCi-2021
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Vasileios Tzortzis, Professor of Urology, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 49616/11.05.2021
Record Dates: First submitted 2021-05-13; First posted 2021-05-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Phimosis; Foreskin; Tightness; Redundant Prepuce
MeSH Terms: conditions — Phimosis | interventions — Circumcision, Male

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Circumcision (Other): Adult patients treated with circumcision
  Interventions: Procedure: Circumcision in adults
- Circumcision with device (Active Comparator): Adult patients treated with sterile single-use circular stapling device CIRCCURERII (Jiangxi Langhe Medical Instrument Co., Ltd., Guangzhou, China)
  Interventions: Device: Circumcision in adults using sterile single-use circular stapling device

INTERVENTIONS:
Device: Circumcision in adults using sterile single-use circular stapling device — Circumcision in adults using sterile single-use circular stapling device CIRCCURER II (Jiangxi Langhe Medical Instrument Co., Ltd., Guangzhou, China)
  Other Names: Sterile single-use circular stapling device
  Arms: Circumcision with device
Procedure: Circumcision in adults — Circumcision in adults
  Other Names: Circumcision
  Arms: Circumcision

SUMMARY:
Evaluation of the safety and efficacy of the sterile single-use circular stapling device CIRCCURER II (Jiangxi Langhe Medical Instrument Co., Ltd., Guangzhou, China) in comparison with circumcision in adults patients with pathological foreskin (phimosis, stenosis, redundant prepuce)

ELIGIBILITY:
Inclusion criteria :phimosis, stenosis of foreskin, redundant prepuce

Exclusion criteria : active inflammation of foreskin

Ages: 16 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Only males suffer from foreskin pathologic conditions
Enrollment: 100 (Estimated)
Dates: Start 2021-05-11 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Bleeding | Intraoperatively
  Number of gauzes used intraoperatively
Postoperative hematoma | First postoperative day
  Measurement defined as follows: mild=1, moderate=2 and large=3, according to the surgeon's estimation
Postoperative hematoma | Seventh postoperative day
  Measurement defined as follows: mild=1, moderate=2 and large=3, according to the surgeon's estimation
Postoperative oedema | Twenty first postoperative day
  Measurement defined as follows: mild=1, moderate=2 and large=3, according to the surgeon's estimation
Duration of procedure | Intraoperative (Measurement begins at the time of the beginning of the sterilisation of the surgical field and ends at the time of the completion of the bandeage of the wound)
  Minutes

SECONDARY OUTCOMES:
Postoperative oedema | First postoperative day
  Measurement defined as follows: mild=1, moderate=2 and large=3, according to the surgeon's estimation
Postoperative oedema | Seventh postoperative day
  Measurement defined as follows: mild=1, moderate=2 and large=3, according to the surgeon's estimation
Aesthetic result | Nineteenth postoperative day
  Visual analogue scale from 0 to 10, as follows: 0 - 5 = unsatisfactory, 6 - 7 = moderately satisfactory, 8 - 9 = very satisfactory, 10 = excellent, according to the patient's estimation

OTHER OUTCOMES:
Pain feeling | Intraoperatively
  Visual analogue scale from 0 to 10, as follows: 0 = no pain, 1-3 = mild pain, 4-6 = moderate pain, 7-9 = very severe pain and 10 = worst possible pain, according to the patient's estimation
Anaesthesia | Immediately preoperatively
  Quantity of applied lidocaine hydrochloride 2% w/v in milliliters
Used sutures | Intraoperatively
  Absolute number of used sutures

CONTACTS AND LOCATIONS:
Overall Officials: Vasileios Tzortzis, Professor, Principal Investigator — Urology Department, University of Thessaly, University Hospital of Larissa, Greece
Locations (1):
- Urology Department, University of Thessaly, University Hospital of Larissa, Larissa, Larissa/Thessaly, Greece

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: After a publication and for a period of 2 years